CLINICAL TRIAL: NCT01836757
Title: The Effect of Methyl-Sulphonyl-Methane on Osteoarthritis and Joint Cartilage Associated With the Degeneration of the Chondrocyte
Brief Title: Effect of Methyl-Sulphonyl-Methane on Osteoarthritis and Cartilage
Acronym: msm
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: G.Papanikolaou Research Group (Other)
Responsible Party: Principal Investigator, Thomas Pagonis, Orthopaedic Surgeon, G.Papanikolaou Research Group
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: msm2012
Record Dates: First submitted 2013-03-13; First posted 2013-04-22 (Estimated); Last update posted 2013-04-22 (Estimated); Status verified 2013-04

CONDITIONS: Osteoarthritis
Keywords: osteoarthritis; CAM treatments; MSM
MeSH Terms: conditions — Osteoarthritis | interventions — dimethyl sulfone

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- MSM group (Experimental): Intervention is MSM 3 gr twice a day for 26 weeks (6 gr/day total)
  Interventions: Drug: MethylSulfonylMethane (MSM)
- Placebo Group (Placebo Comparator): Placebo 3 gr twice a day for 26 weeks (6 gr/day total)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: MethylSulfonylMethane (MSM) — Intervention is MSM 3 gr twice a day for 26 weeks (6 gr/day total)
  Arms: MSM group
Drug: Placebo
  Arms: Placebo Group

SUMMARY:
To delineate the effect of MSM on osteoarthritis

DETAILED DESCRIPTION:
Objective: To delineate the effect of MSM on osteoarthritis of large joints. Design: Randomized, double-blind, placebo-controlled trial including an intervention and a placebo group. One hundred men and women, with hip and/or knee OA to be divided in 2 groups. Intervention is either MSM 3 gr twice a day for 26 weeks (6 gr/day total) for one group and placebo for the other. Outcomes measured are the Western Ontario and McMaster University Osteoarthritis Index visual analogue scale (WOMAC), patient and physician assessments and SF-36 (overall health-related quality of life).

ELIGIBILITY:
Inclusion Criteria:

* Knee and hip OA
* men and women >45 years of age

Exclusion Criteria:

* any other type of arthritis
* chronic pain syndrome
* arthroscopic surgery in the past 8 months
* intra-articular corticosteroidsin the past 8 months
* hyaluronic acid injections in the past 8 months
* narcotic pain killers use
* renal or hepatic disease
* body mass index (BMI) >45 kg/m2
* cancer

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2012-09; Primary Completion 2013-09 (Estimated); Study Completion 2013-10 (Estimated)

PRIMARY OUTCOMES:
Number of participants with improved Mobility | 26 weeks
  Randomized, double-blind, placebo-controlled trial including an intervention and a placebo group. One hundred men and women, with hip and/or knee OA were divided in 2 groups. Intervention was either MSM 3 gr twice a day for 26 weeks (6 gr/day total) for one group and placebo for the other. Outcomes measured were the Western Ontario and McMaster University Osteoarthritis Index visual analogue scale (WOMAC)

SECONDARY OUTCOMES:
Pain Scores on the Visual Analog Scale | 26 weeks
  On the same two groups (MSM and Placebo)we measured the improvement of quality of life through pain relief as measured by use of SF-36 (overall health-related quality of life)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Pagonis, MD, PhD, Principal Investigator — Aristotle's University of Thessaloniki
Locations (1):
- G. Papanikolaou Hospital, Thessaloniki, Thessaloniki, Greece